CLINICAL TRIAL: NCT03240744
Title: Study on Immunogenicity of Inactivated Enterovirus 71 (EV71) Vaccine (Human Diploid Cell, KMB-17) in Large-scale Healthy Children in China
Brief Title: The Phase IVc of Inactivated Enterovirus 71 Vaccine (Human Diploid Cell)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, Qihan Li, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-003-02
Record Dates: First submitted 2017-06-22; First posted 2017-08-07 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-04

CONDITIONS: Hand, Foot and Mouth Disease (HFMD)
Keywords: immunogenicity; safety; Hand, Foot and Mouth Disease (HFMD)
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Intervention Model Description: Inactivated EV71 vaccine (KMB-17 cells)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaccine (3.0EU) (Experimental): healthy children (6-71 months old) have been injected by inactivated EV71 vaccine (KMB-17) of 3.0 EU (neutralization antibodies titer unit; 100 U in phase III clinical trials, or 320 EU (Elisa assay unit) in phase I and II clinical trials)
  Interventions: Biological: Inactivated EV71 vaccine (human diploid cell, KMB-17)

INTERVENTIONS:
Biological: Inactivated EV71 vaccine (human diploid cell, KMB-17) — 3.0 EU of inactivated enterovirus 71 vaccine (KMB-17) on day 0, 28.

SUMMARY:
Enterovirus 71 (EV71), a major pathogen causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Its infection occasionally leads to severe diseases and death, with central nervous system (CNS) damage.

Recently, except of inactivated vaccine, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, such as attenuated vaccine, subunit vaccine. A formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been finished phase I, II and III clinical trials and licensed by SFDA in China at Dec. 3, 2015. Based on the results of clinical trials, the protective efficacy of inactivated EV71 vaccine is 97% against HFMD caused by EV71. The phase IV clinical trial has been carried out from July 2016. The purpose of phase IVc is to evaluated the immunogenicity of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old) in Hubei Province, China.

DETAILED DESCRIPTION:
There are two parts of phase IVc clinical trials have been performed. First, to evaluate the immunogenicity of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old), within 56-day-post-immunized.

Second, to long-term immunogenicity of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (6-71 months old children) as established by medical history and clinical examination
* The subjects' legal guardian must be aware of this vaccines
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0 ℃
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol
* Persist for a 14-month visit (and receive blood, stool (or specimens by means of a swab) tests according to program requirements in immunogenicity observation group)

Exclusion Criteria:

* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 15 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Fever before vaccination, axillary temperature ﹥37.0 ℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140 mmHg and/ or diastolic blood pressure ﹥90 mmHg; systolic blood pressure ﹤90 mmHg and/or diastolic blood pressure ﹤60 mmHg
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives
* take part into other vaccine or drug clinical trials in last half year

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of children | at 28 days after finishing 2 doses immunization
  Bloods were obtained at 0 and 56 days after first vaccination. The antibody titers were tested in serum of children. And the seroconversion rate of anti-EV71 antibodies was calculated.
Evaluate the antibody titers of anti-EV71 antibodies in serum of children | at 28 days after finishing 2 doses immunization
  Bloods were obtained at 0 and 56 days after first vaccination. The antibody titers were tested in serum of children. And the seroconversion rate of anti-EV71 antibodies was calculated.

SECONDARY OUTCOMES:
Evaluate long-term of the seroconversion rate of anti-EV71 antibodies in serum of children | Up to 3 years after finishing 2 doses immunization
  Bloods were obtained at 0, 28 and 56 days after first vaccination, and 180, 360 and 720 days after 2 doses immunization. The antibody titers were tested in serum of children. And the seroconversion rate of anti-EV71 antibodies was calculated.
Evaluate long-term of the antibody titers of anti-EV71 antibodies in serum of children | Up to 3 years after finishing 2 doses immunization
  Bloods were obtained at 0, 28 and 56 days after first vaccination, and 180, 360 and 720 days after 2 doses immunization. The antibody titers were tested in serum of children. And the seroconversion rate of anti-EV71 antibodies was calculated.

OTHER OUTCOMES:
Incidence of treatment adverse events | Up to 3 years after finishing 2 doses immunization
  The adverse events were observed and recorded within 30 minutes post immunization (p.i.), within 0-1 days post immunization (d.p.i.), within 1-3 d.p.i. and within 3-7 d.p.i. after the 1st injection, as well as after the 2nd injection. And the adverse events were also observed and recorded following within 3 years after finishing 2 doses immunization.

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Guan, M.S., Principal Investigator — Hubei Province Center for Diseases Control and Prevention
Locations (1):
- Hubei Province Center for Diseases Control and Prevention, Wuhan, Hubei, China